CLINICAL TRIAL: NCT01838148
Title: BASEL VIII Trial - Biochemical and Electrocardiographic Signatures in the Detection of Exercise-induced Myocardial Ischemia
Brief Title: Biochemical and Electrocardiographic Signatures in the Detection of Exercise-induced Myocardial Ischemia
Acronym: BASEL VIII
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: BASEL VIII
Record Dates: First submitted 2013-04-12; First posted 2013-04-23 (Estimated); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease; Angina, Stable; Exercise Test; Biological Markers; SPECT
Keywords: coronary artery disease; angina, stable; exercise test; biological Markers; SPECT
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA, plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary aim is to perform the largest study worldwide to evaluate novel biochemical and electrocardiographic signatures alone as well as in combination with the standard 12-lead exercise ECG in the detection of exercise-induced myocardial ischemia (diagnostic endpoint). The secondary aim is to evaluate these innovative tools in the risk prediction for the occurrence of cardiovascular death and acute myocardial infarction during long-term follow-up.

DETAILED DESCRIPTION:
Background: The detection of coronary artery disease (CAD) is one of the most important tasks in medicine. Exercise-induced myocardial ischemia is the pathophysiological hallmark of stable CAD. Currently, sophisticated imaging techniques including coronary angiography, rest/stress myocardial perfusion single-photon emission computed tomography (SPECT), and coronary CT-scanning are required to accurately detect CAD. Unfortunately, these techniques are associated with inherent risks due to substantial radiation exposure, intraarterial or intravenous application of iodinated contrast media, mechanical complications, require referral to a specialist, and are very costly. In addition, most of them provide anatomical but not functional information. For clinical practice, functional information that differentiates lesions that cause exercise-induced myocardial ischemia from functionally irrelevant lesions is critical. Exercise electrocardiography (ECG) is a widely used simple and non-invasive functional test, which however has imperfect sensitivity and specificity (both below 75%) in the detection of CAD. Novel cardiac biomarkers as well as novel computer-based quantitative approaches to analyse the ECG signal recorded during exercise offered by advances in information technology and signal processing may provide incremental value to the exercise ECG and thereby improve clinical care.

Aim: The primary aim is to perform the largest study worldwide to evaluate novel biochemical and electrocardiographic signatures alone as well as in combination with the standard 12-lead exercise ECG in the detection of exercise-induced myocardial ischemia (diagnostic endpoint). The secondary aim is to evaluate these innovative tools in the risk prediction for the occurrence of cardiovascular death and acute myocardial infarction during long-term follow-up.

Methodology: We will enroll approximately 4200 consecutive patients with suspected exercise induced myocardial ischemia referred for rest/ergometry myocardial perfusion SPECT. SPECT findings (complemented by coronary angiography and fractional flow reserve [FFR, if availabe] findings in patients who obtain both investigations) are used to adjudicate and quantify the presence of myocardial ischemia (the primary diagnostic end point). Clinical long-term follow-up will be obtained at 1 year, 2 years, 5 years and 8 years to record death, cardiovascular death, and acute myocardial infarction as well as coronary revascularisation.

Investigational tests: Venous blood samples will be collected before exercise stress testing for the determination of biochemical signatures possibly associated with myocardial ischemia including high-sensitivity cardiac troponin I, high-sensitivity cardiac troponin T, B-type natriuretic peptide, IL-6, and cardiac microRNA. In addition, continuous ECG signals are recorded using 12 leads (16 leads in a subset of patients) and 24-bit amplitude resolution with 8000 Hz sampling frequency before, during and after the stress test. Novel methods of computer-based ECG signal-processing technology will be used to decipher electronic markers of myocardial ischemia and to develop improved software algorithms for automated ECG interpretation. All investigational tests will be performed in a blinded fashion.

Potential Significance: We hypothesize that biochemical and electrocardiographic signals of myocardial ischemia will significantly improve the non-invasive detection of exercise-induced myocardial ischemia. This would markedly improve the initiation of treatment in affected patients and thus advance medical management of patients with suspected CAD. In addition, this approach would help to simplify (exercise ECG versus myocardial SPECT) the non-invasive detection of exercise-induced myocardial ischemia and help to avoid the inherent health hazards associated current radiologic imaging procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with suspected exercise-induced myocardial ischemia referred for rest/ergometry myocardial perfusion SPECT

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Unable or unwilling to give informed consent
* Symptoms at rest or minor exertion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients presenting with suspected exercise-induced myocardial ischemia referred for rest/ergometry myocardial perfusion SPECT.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2004-05; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic utility of novel biochemical and electrocardiographic signatures | baseline
  Diagnostic utility of biochemical (i.e. cardiac troponin, brain natriuretic peptide) and electrocardiographic signatures alone as well as in combination with the standard 12-lead exercise ECG in the detection of exercise-induced myocardial ischemia, mainly quantified by the area under the receiver operating characteristics curves (AUC ROC) and positive/negative predictive values, respectively.

SECONDARY OUTCOMES:
One year event-free survival | 360 days
  Prognostic utility of biochemical (i.e. cardiac troponins, brain natriuretic peptides) and electrocardiographic signatures in the risk prediction for the occurrence of cardiovascular death and acute myocardial infarction
Two year event-free survival | 2 years
  Prognostic utility of biochemical (i.e. cardiac troponins, brain natriuretic peptides) and electrocardiographic signatures in the risk prediction for the occurrence of cardiovascular death and acute myocardial infarction
Five year event-free survival | 5 years
  Prognostic utility of biochemical (i.e. cardiac troponins, brain natriuretic peptides) and electrocardiographic signatures in the risk prediction for the occurrence of cardiovascular death and acute myocardial infarction
Eight year event-free survival | 8 years
  Prognostic utility of biochemical (i.e. cardiac troponins, brain natriuretic peptides) and electrocardiographic signatures in the risk prediction for the occurrence of cardiovascular death and acute myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mueller, Prof. Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Amrein M, Li XS, Walter J, Wang Z, Zimmermann T, Strebel I, Honegger U, Leu K, Schafer I, Twerenbold R, Puelacher C, Glarner N, Nestelberger T, Koechlin L, Ceresa B, Haaf P, Bakula A, Zellweger M, Hazen SL, Mueller C. Gut microbiota-dependent metabolite trimethylamine N-oxide (TMAO) and cardiovascular risk in patients with suspected functionally relevant coronary artery disease (fCAD). Clin Res Cardiol. 2022 Jun;111(6):692-704. doi: 10.1007/s00392-022-01992-6. Epub 2022 Feb 26. PMID 35220448
- [Derived] Walter JE, Amrein MLF, Schafer I, Zimmermann T, Lopez-Ayala P, Boeddinghaus J, Twerenbold R, Puelacher C, Nestelberger T, Wussler D, Honegger U, Badertscher P, Eugen-Olsen J, Koechlin L, Fahrni G, Jeger R, Kaiser C, Zellweger M, Mueller C. Soluble urokinase plasminogen activator receptor and functionally relevant coronary artery disease: a prospective cohort study. Biomarkers. 2022 May;27(3):278-285. doi: 10.1080/1354750X.2022.2038269. Epub 2022 Feb 15. PMID 35112976
- [Derived] Walter J, du Fay de Lavallaz J, Koechlin L, Zimmermann T, Boeddinghaus J, Honegger U, Strebel I, Twerenbold R, Amrein M, Nestelberger T, Wussler D, Puelacher C, Badertscher P, Zellweger M, Fahrni G, Jeger R, Kaiser C, Reichlin T, Mueller C. Using High-Sensitivity Cardiac Troponin for the Exclusion of Inducible Myocardial Ischemia in Symptomatic Patients: A Cohort Study. Ann Intern Med. 2020 Feb 4;172(3):175-185. doi: 10.7326/M19-0080. Epub 2020 Jan 7. PMID 31905377
- [Derived] Badertscher P, Strebel I, Honegger U, Schaerli N, Mueller D, Puelacher C, Wagener M, Abacherli R, Walter J, Sabti Z, Sazgary L, Marbot S, du Fay de Lavallaz J, Twerenbold R, Boeddinghaus J, Nestelberger T, Kozhuharov N, Breidthardt T, Shrestha S, Flores D, Schumacher C, Wild D, Osswald S, Zellweger MJ, Mueller C, Reichlin T. Automatically computed ECG algorithm for the quantification of myocardial scar and the prediction of mortality. Clin Res Cardiol. 2018 Sep;107(9):824-835. doi: 10.1007/s00392-018-1253-z. Epub 2018 Apr 17. PMID 29667014
- [Derived] Puelacher C, Wagener M, Honegger U, Assadian M, Schaerli N, Mueller D, Strebel I, Twerenbold R, Boeddinghaus J, Nestelberger T, Wildi K, Sabti Z, Sazgary L, Badertscher P, du Fay de Lavallaz J, Marbot S, Kaiser C, Wild D, Zellweger MJ, Reichlin T, Mueller C. Combining high-sensitivity cardiac troponin and B-type natriuretic peptide in the detection of inducible myocardial ischemia. Clin Biochem. 2018 Feb;52:33-40. doi: 10.1016/j.clinbiochem.2017.10.014. Epub 2017 Nov 8. PMID 29107010
- [Derived] Sou SM, Puelacher C, Twerenbold R, Wagener M, Honegger U, Reichlin T, Schaerli N, Pretre G, Abacherli R, Jaeger C, Rubini Gimenez M, Wild D, Rentsch KM, Zellweger MJ, Mueller C. Direct comparison of cardiac troponin I and cardiac troponin T in the detection of exercise-induced myocardial ischemia. Clin Biochem. 2016 Apr;49(6):421-432. doi: 10.1016/j.clinbiochem.2015.12.005. Epub 2015 Dec 17. PMID 26708172